CLINICAL TRIAL: NCT00136097
Title: Study on the Infection Risk of Long Dwell Period Catheters in High Risk ICU Patients
Brief Title: Study on the Infection Risk of Long Dwell Period Catheters in High Risk Intensive Care Unit (ICU) Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2004/266
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Burns
Keywords: colonisation of the catheter
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Placement of a silver impregnated central venous catheter

SUMMARY:
This is an evaluation of the use of silver impregnated catheters in burn patients to reduce catheter colonisation compared to the standard central venous catheter without antiseptic activity.

ELIGIBILITY:
Inclusion Criteria:

* Burn patient
* Placement of a new trilumen central venous catheter

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142
Dates: Start 2005-08; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Degree of colonisation of the central venous catheter at the moment of removal

SECONDARY OUTCOMES:
Incidence of a catheter related blood stream infection during the presence of the catheter

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Colpaert, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be